CLINICAL TRIAL: NCT06102785
Title: Phase II Clinical Study of Fruquintinib Combined TAS102 for Second-line Treatment of Advanced Gastric Cancer
Brief Title: Fruquintinib Combined With TAS102 for Advanced Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJMUCH-GI-GC06
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; second-line treatment; Fruquintinib; TAS102
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; trifluridine tipiracil drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fruquintinib combined with TAS102: Fruquintinib 4mg d1-21, q4w TAS102 35mg/m2，bid，d1-5，d15-19，q4w
  Interventions: Drug: Fruquintinib, TAS102

INTERVENTIONS:
Drug: Fruquintinib, TAS102 — Fruquintinib combined with TAS102

SUMMARY:
This is a prospective, single-center, open, single-arm clinical study to observe and evaluate the efficacy and safety of Fruquintinib combined with TAS102 for second-line treatment of advanced gastric cancer.

DETAILED DESCRIPTION:
A prospective study of Fruquintinib combined with TAS-102 for the posterior line treatment of advanced colorectal cancer is ongoing (NCT05004831). Both Fuquinitinib and TAS-102 are oral drugs, which are convenient to use and avoid the burden of frequent hospitalization. Whether this combination has considerable efficacy in gastric cancer is not clear.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. The ECOG score is 0-1 and does not deteriorate within 7 days.
3. Patients with histologically confirmed, metastatic, or unresectable locally advanced gastric cancer or GEJ adenocarcinoma.
4. Previously received one systemic chemotherapy regimen for this cancer and progressed; Or have received adjuvant chemotherapy, but have disease progression or recurrence within 6 months after the end of treatment.
5. Measurable lesions that meet RECIST 1.1 criteria.
6. Have adequate organ and bone marrow function, laboratory tests meet the following requirements:

   1. HGB≥90g/L;
   2. NEUT≥1.5×10^9/L;
   3. PLT ≥80×10^9/L;
   4. TBIL≤1.5 times upper limit of normal value (ULN);
   5. ALT and AST≤2.5 x ULN; In liver metastasis, ALT and AST≤5×ULN;
   6. Endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula);
   7. Urinary protein < (++), or 24-hour urinary protein volume < 1.0 g.
7. Normal coagulation function, no active bleeding

   1. International standardized ratio INR≤1.5;
   2. Partial thromboplastin time APTT≤1.5 ULN.
8. Women of childbearing age must undergo a negative pregnancy test (serum or urine) within 14 days prior to enrollment and voluntarily use an appropriate method of contraception during the observation period and within 8 weeks after the last dose of the study drug; For men, they should be surgically sterilized or consent to an appropriate method of contraception during the observation period and for 8 weeks after the last administration of the study drug.
9. Expected survival ≥3 months.
10. Patients voluntarily joined the study and signed an informed consent form (ICF).
11. It is expected that the compliance is good, and the efficacy and adverse reactions can be followed up according to the protocol requirements.

Exclusion Criteria:

1. Previous treatment with VEGFR inhibitors;
2. Previously received paclitaxel therapy (except for those who received paclitaxel therapy in neoadjuvant or adjuvant therapy, and the treatment ended more than 6 months after the disease progression);
3. Receive live vaccine within 4 weeks prior to enrollment or possibly during the study period;
4. Had active autoimmune disease or history of autoimmune disease within 4 weeks prior to enrollment;
5. Previously received allogeneic bone marrow transplantation or organ transplantation;
6. Hypertension that could not be controlled by drugs before enrollment was defined as: systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥90 mmHg;
7. Had any disease or condition affecting drug absorption before enrollment, or the patient could not take drugs orally;
8. Gastrointestinal diseases such as active ulcer of stomach and duodenum, ulcerative colitis, or active bleeding of unexcised tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers before enrollment;
9. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months > 30 mL, hematemesis, stool, stool blood), hemoptysis, or thromboembolic events (including stroke events and/or transient ischemic attacks) within 12 months;
10. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure > Level 2; Ventricular arrhythmias requiring medical treatment; LVEF (Left ventricular Ejection Fraction) < 50%;
11. Active or uncontrolled severe infection (≥CTCAE v5.0 grade 2 infection);
12. Known human immunodeficiency virus (HIV) infection. Known history of clinically significant liver disease, including viral hepatitis [Known hepatitis B virus (HBV) carriers must rule out active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or > 2000 IU/ mL); known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL);
13. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, reasonably suspects that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk;
14. The patients considered by the investigators to be unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced gastric cancer with second-line treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Time from the start of treatment to the progression of the disease

SECONDARY OUTCOMES:
Disease Control rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The proportion of CR,PR and SD
The Overall Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The proportion of CR and PR
Overall survival | From date of randomization until the date of death from any cause or the last visit date, whichever came first, assessed up to 60 months
  Time from the start of treatment to the occurrence of death

CONTACTS AND LOCATIONS:
Overall Officials: Ting Deng, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Zhang Y, Wang ZX, Shen L, et al. A phase Ib/II study of fruquintinib in combination withpaclitaxel as the second-line therapy for advanced gastric cancer. Cancer Commun (Lond) 2023; 43:150-153. 2. Shitara K, Doi T, Dvorkin M, et al. Trifluridine/tipiracil versus placebo in patients with heavilypretreated metastatic gastric cancer (TAGS): a randomised, double-blind, placebo-controlled, phase 3trial. Lancet Oncol 2018; 19: 1437-1448. 3. Gou M, Qian N, Zhang Y, et al. Fruquintinib in Combination With PD-1 Inhibitors in PatientsWith Refractory Non-MSI-H/pMMR Metastatic Colorectal Cancer: A Real-World Study in China. FrontOncol 2022; 12: 851756. 4. Takahara Y, Tanaka T, Ishige Y, et al. Efficacy and predictors of rechallenge with immunecheckpoint inhibitors in non-small cell lung cancer. Thorac Cancer 2022; 13: 624-630. 5. Nukatsuka M, Fujioka A, Nagase H, et al. Evaluation of a novel combination therapy, basedon trifluridine/tipiracil and fruquintinib, against colorectal cancer. Chemotherapy 2023.